CLINICAL TRIAL: NCT02441777
Title: Polarization Sensitive Optical Coherence Tomography (PS-OCT) for Retinal Imaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Benjamin Vakoc, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014P001042
Record Dates: First submitted 2015-04-27; First posted 2015-05-12 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: retinal imaging; optical imaging; optical coherence tomography; polarization sensitive coherence tomography
MeSH Terms: interventions — Optical Imaging; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Control: Healthy (Experimental): Polarization Sensitive Optical Coherence Tomography (PS-OCT) Imaging will be used to look at the nerve fiber layer (NFL) in the healthy retina.
  Interventions: Device: Polarization-Sensitive OFDI

INTERVENTIONS:
Device: Polarization-Sensitive OFDI — OCT Imaging of the eye
  Other Names: Optical Imaging; Optical Coherence Tomography; OCT; Optical Frequency Domain Imaging

SUMMARY:
The aim of this pilot study is to assess the ability of a new polarization sensitive optical coherence tomography system to obtain high-quality images of retinal birefringence.

DETAILED DESCRIPTION:
Glaucoma is the second leading cause of blindness in the world. The current clinical standard-of-care procedure to diagnose glaucoma is visual field testing with disc photography. Visual field testing is subjective both in the patient's feedback and the physician's interpretation of this feedback, and disc photography requires a physician's subjective interpretation. As a result, it is estimated that current methods can diagnose glaucoma only after 40% of the nerve fiber layer (NFL) has been lost. Since glaucoma leads to significant changes in both NFL thickness and NFL optical birefringence, non-invasive imaging of these properties could potentially enable diagnosis of glaucoma prior to changes in vision. Optical Coherence Tomography (OCT) is routinely used in retinal imaging, and its ability to detect changes in NFL health is being actively studied. To detect NFL optical birefringence, a specialized variation of OCT termed polarization sensitive OCT (PS-OCT) is required. Because of high noise in PS-OCT images, prior studies have been unable to detect NFL changes in birefringence.

We have recently developed new methods for performing highly sensitive polarization-sensitive OCT. These changes are algorithmic in nature, and use the same optical wavelengths and powers as clinically deployed OCT retinal imaging instruments. In benchtop studies, these algorithmic changes improve the signal-to-noise ratio (SNR) of PS-OCT images. We propose to conduct a pilot study in normal, healthy subjects to evaluate if these changes improve the SNR of NFL birefringence images.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 18-85 years
2. Healthy normal subjects with no significant eye disease, except for mild cataracts
3. Subjects with clear enough cornea or clear enough media to permit imaging
4. Subjects with refractive error between -5.00 sph to +5.00 sph

Exclusion Criteria:

1. Subjects who have occludable narrow angles (without a patent peripheral iridotomy) or any other ocular or systemic pathology, which precludes safe dilation
2. Subjects whose eyes have been dilated for over 6 hours will not be eligible for imaging.
3. Subjects who do not or cannot understand the instructions for the PS-OCT imaging
4. Subjects who are pregnant and/or breastfeeding. Date of last menstrual cycle will also be included.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Average nerve fiber layer (NFL) birefringence | At time of imaging
  Measured birefringence values will be compared to normative values from literature

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Vakoc, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States